CLINICAL TRIAL: NCT02752880
Title: The Efficacy and Safety of Concentrated Herbal Extract Granules, YH1, as an Add-On Medication in Poorly Controlled Type 2 Diabetes: A Randomized, Double-Blind, Placebo-Controlled Pilot Trial
Brief Title: YH1 in Poorly Controlled Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-7934A3,105-7009C,106-0917C
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Coptidis rhizoma extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- YH1 group (Experimental): YH1 with one batch number was manufactured by Sun Ten Pharmaceutical Co., Ltd., a renowned manufacturer of concentrated herbal extract granules conforming to the standards of good manufacturing practices (GMP) in New Taipei City, Taiwan. YH1 contains Rhizoma Coptidis (50 %) and Shen-Ling-Bai-Zhu-San (SLBZS) (50 %). SLBZS consists of Radix Ginseng, Poria, Rhizoma Atractylodis macrocephalae, Semen Lablab album, Rhizoma Dioscoreae, Embryo Nelumbinis, Radix Platycodonis, Semen Coicis, Fructus Amomi, Fructus Jujubae, and Radix Glycyrrhizae at a 3:3:3:2.3:3:1.5:1.5:1.5:1.5:1.5:3 ratio. Subjects in the YH1 group orally ingested two packages of granules (3 g/package) three times daily with warm water after a meal for 12 consecutive weeks.
  Interventions: Drug: YH1 group
- placebo group (Placebo Comparator): The placebo was also prepared as granules by Sun Ten Pharmaceutical Co., Ltd., and the packaging of the placebo was identical to that of YH1. Subjects in the placebo group orally ingested two packages of granules (3 g/package) three times daily with warm water after a meal for 12 consecutive weeks.
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: YH1 group — Participants were randomly assigned 1:1 to receive either YH1 or placebo for 12 consecutive weeks.
  Other Names: Rhizoma Coptidis and Shen-Ling-Bai-Zhu-San
  Arms: YH1 group
Drug: placebo group — Participants were randomly assigned 1:1 to receive either YH1 or placebo for 12 consecutive weeks.
  Arms: placebo group

SUMMARY:
Type 2 diabetes mellitus is a chronic metabolic disease that seriously affects patients worldwide, and it is always among the top 10 causes of death in Taiwan. To date, still many patients who take more than three kinds of oral hypoglycemic agents could not effectively control their glycohemoglobin levels in clinics. Hypoglycemia as well as weight gain are common side effect with insulin therapy, and many patients in Taiwan are not willing to receive insulin injection. It is common for diabetic patients treated with Chinese herbal medicine in China currently, and some therapeutic effects have been published in international journals. In this study, we will evaluate whether Chinese herbal medicine, YH1, enhances the glycemic control and is safe as add-on medication in poorly controlled type 2 diabetes patients.

A total of 46 poorly controlled type 2 diabetes patients with glycohemoglobin ≥ 7% from Endocrinology and Metabolism clinics or Internal Chinese Medicine clinics will be enrolled in this randomized double-blind placebo-controlled trial. Subjects will be randomly assigned to receive either YH1 (6 g) or the placebo three times per day for 12 consecutive weeks. All subjects in both groups will also continuously receive their oral hypoglycemic agents without any dose or medicine change. During this 12-week period, the glycohemoglobin, fasting plasma glucose, 2h postprandial glucose, waist circumference, body weight, and body mass index will be assessed. In addition, insulin resistance, β -cell function, lipid profile, liver and renal function will also be evaluated. Independent statisticians will perform the data analysis at the end of the trial.

DETAILED DESCRIPTION:
The YH1 in one batch number was used, manufactured by Sun Ten Pharmaceutical Co., LTD., a renowned GMP manufacturer of concentrated herbal extract granules conforming to international standards. The YH1 was prepared in small granules, including concentrated herbal extract granules of Rhizoma Coptidis (50%) and SLBZS (50%). Both medicines have already been approved by the Ministry of Health and Welfare in Taiwan as ethical drugs. YH1 granules were packed in aluminum foil packages. The placebo was also prepared as granules by Sun Ten Pharmaceutical Co., LTD., and the packaging of the placebo was identical to that of YH1. The chemical composition of YH1 was analyzed and profiled by using a high performance liquid chromatography (HPLC) with photodiode array (PDA) detection. Fourteen components, allantoin, atractylenolide III, berberine, coptisine, ginsenoside Rb1, ginsenoside Re, ginsenoside Rg1, glycyrrhizin, liquiritin, pachymic acid, palmatine, platycodin D, magnoflorin and quercitrin, were simultaneously used in the qualitative analysis under the developed HPLC-PDA method. As for the quantitative detection, each gram of YH1 contained 20.05 mg berberine.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75 years of age;
2. Diagnosed as type 2 diabetics based on World Health Organization criteria [1];
3. Body mass index (BMI) ≥ 23 kg/m2;
4. Have been treated with ≥ 3 kinds of oral hypoglycemic agents (OHAs) with persistent (> 6 months) high HbA1c (≥ 7.0 %).

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, or other specific types of diabetes;
2. Have received insulin therapy in the past three months;
3. Have serious gastrointestinal (GI) tract diseases, such as peptic ulcers or GI tract bleeding;
4. Experience stressful situations, including diabetic ketoacidosis, nonketotic hyperosmolar diabetic coma, severe infection, or surgery in the previous one month;
5. Suffer from hepatic insufficiency with alanine aminotransferase (ALT) 2 times the upper limit of normal or renal insufficiency with estimated glomerular filtration rate (eGFR) < 60;
6. Uncontrolled hypertension (blood pressure ≥ 160/100 mmHg);
7. Mental illness, abused or addicted to alcohol, psychoactive substances or other drugs;
8. Pregnant, lactating, or plan to become pregnant;
9. Hemoglobin disease or chronic anemia;
10. Have underlying conditions that could lead to poor compliance;
11. History of cerebrovascular disease or myocardial infarction;
12. Have undergone Chinese medicine treatment in the past two weeks.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsiang Huang, MD, Principal Investigator — Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Taoyuan District, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- YH1 Three Times Per Day for 12 Consecutive Weeks: The YH1 in one batch number was used, manufactured by a renowned GMP manufacturer of concentrated herbal extracts conforming to international standards.
- Placebo: placebo three times per day for 12 consecutive weeks.
  placebo
Period: Overall Study
Arm/Group | YH1 Three Times Per Day for 12 Consecutive Weeks | Placebo
Started | 23 | 23
Completed | 21 | 20
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- YH1 Group: YH1 three times per day for 12 consecutive weeks.
- Placebo Group: placebo three times per day for 12 consecutive weeks.
- Total: Total of all reporting groups
Arm/Group | YH1 Group | Placebo Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Median (Full Range); unit: years] | 50 [33 to 69] | 56 [40 to 66] | 52 [33 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 8 | 12 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 20 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HbA1c [Median (Full Range); unit: %] | 8.1 [7.5 to 11.3] | 8.7 [7.6 to 11.8] | 8.6 [7.5 to 11.8]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in HbA1c Level From Baseline to 12 Weeks
Description: The primary efﬁcacy endpoint was the percentage change in HbA1c levels from baseline to 12 weeks. The HbA1c level was measured by HPLC in the Department of Laboratory Medicine at Chang Gung Memorial Hospital.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: percentage change
Arm/Group | YH1 Group | Placebo Group
Number analyzed (Participants) | 21 | 20
percentage change | -11.1 [-30.2 to 14.1] | 0.0 [-20.4 to 7.3]

2. Secondary Outcome: The Percentage Change in 2hPG From Baseline to Week 12
Description: The secondary efﬁcacy endpoint was the percentage change in 2hPG level from baseline to 12 weeks by using enzymatic method in the Department of Laboratory Medicine at Chang Gung Memorial Hospital.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: percentage change
Groups:
- Placebo: placebo three times per day for 12 consecutive weeks.
Arm/Group | YH1 Group | Placebo
Number analyzed (Participants) | 21 | 20
percentage change | -26.2 [-60.3 to 94.1] | 5.1 [-43.0 to 90.6]

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- YH1 Group: During 12 weeks of YH1 treatment, participants were encouraged to report any discomfort to the project manager throughout the trial. Adverse events including any undesirable or unintended symptoms were assessed regardless of the causal relationship with the study drug.
- Placebo Group: During 12 weeks of placebo treatment, participants were encouraged to report any discomfort to the project manager throughout the trial. Adverse events including any undesirable or unintended symptoms were assessed regardless of the causal relationship with the study drug.
Arm/Group | YH1 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 12/23 | 13/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YH1 Group (N=23) | Placebo Group (N=23)
abdominal fullness (Gastrointestinal disorders) | 3 | 3
diarrhea (Gastrointestinal disorders) | 7 | 3
dizziness (General disorders) | 0 | 4
upper respiratory tract infection (Infections and infestations) | 4 | 3
nausea (Gastrointestinal disorders) | 3 | 2
acid reflux (Gastrointestinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT02752880/Prot_SAP_000.pdf